CLINICAL TRIAL: NCT04158687
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of CTP-692 as an Adjunctive Treatment in Adult Patients With Schizophrenia
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of CTP-692 as an Adjunctive Treatment in Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP692.2001
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received CTP-692 matched-placebo powder for oral solution, once daily (QD) for up to 12 weeks.
  Interventions: Drug: Placebo
- CTP-692 1 gram QD (Experimental): Participants received CTP-692 1 gram powder for oral solution, QD for up to 12 weeks.
  Interventions: Drug: CTP-692
- CTP-692 2 grams QD (Experimental): Participants received CTP-692 2 grams powder for oral solution, QD for up to 12 weeks.
  Interventions: Drug: CTP-692
- CTP-692 4 grams QD (Experimental): Participants received CTP-692 4 grams powder for oral solution, QD for up to 12 weeks.
  Interventions: Drug: CTP-692

INTERVENTIONS:
Drug: CTP-692 — Administered as powder for oral solution.
  Arms: CTP-692 1 gram QD; CTP-692 2 grams QD; CTP-692 4 grams QD
Drug: Placebo — Administered as powder for oral solution.
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety and efficacy of 3 different doses of CTP-692 administered once daily (QD) for 12 weeks to adult participants with schizophrenia on stable dopaminergic antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed diagnostic and statistical manual-version 5 (DSM-V5) diagnosis of schizophrenia for the past 2 years
* Patients with clinically stable schizophrenia with residual symptoms defined as positive and negative syndrome scale (PANSS) total score of 70-110
* Patients currently treated with one antipsychotic medication

Exclusion Criteria:

* Patients who, in the opinion of the Investigator, have a history of antipsychotic treatment resistance
* Patients currently taking clozapine
* History of meeting DSM-V5 criteria for moderate to severe alcohol or substance use disorder (other than nicotine or caffeine) within the 6 months before the first Screening Visit
* Patients with positive blood screen for human immunodeficiency virus (HIV) antibody and/or hepatitis B virus surface antigen
* Patients with history of renal disease or those taking medications to treat renal disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Synexus Clinical Research US, Inc., Cerritos, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Pillar Clinical Research, LLC, Lincolnwood, Illinois
  - CBH Health, LLC, Gaithersburg, Maryland
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Synexus Clinical Research US, Inc., Jamaica, New York
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Donald J. Garcia Jr., MD, PA, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in the United States from 26 November 2019 to 22 December 2020.
Pre-assignment Details: 521 participants were screened, out of which 326 participants with schizophrenia who were on a stable dopaminergic antipsychotic medication were enrolled and randomized.
Period: Overall Study
Arm/Group | Placebo | CTP-692 1 Gram QD | CTP-692 2 Grams QD | CTP-692 4 Grams QD
Started | 81 | 81 | 85 | 79
Safety Population (Safety population included all participants who received at least one dose of study medication.) | 81 | 81 | 85 | 78
Efficacy Population (Efficacy population included all participants who received the study medication and had at least one available post-baseline Positive and Negative Syndrome Scale (PANSS) assessment.) | 80 | 81 | 83 | 77
Completed | 64 | 54 | 65 | 66
Not Completed | 17 | 27 | 20 | 13
Not completed — Adverse Event | 2 | 3 | 0 | 3
Not completed — Lost to Follow-up | 5 | 12 | 4 | 5
Not completed — Coronavirus Disease 2019 (COVID-19) Related Reasons | 2 | 3 | 2 | 0
Not completed — Non-Compliance with Study Medication | 2 | 2 | 3 | 0
Not completed — Investigator Decision | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 1 | 0
Not completed — Withdrawal of Consent by Subject | 3 | 3 | 4 | 1
Not completed — Reason not Specified | 3 | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study medication.
Groups:
- Placebo: Participants received CTP-692 matched placebo powder for oral solution, QD for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | CTP-692 1 Gram QD | CTP-692 2 Grams QD | CTP-692 4 Grams QD | Total
Number analyzed (Participants) | 81 | 81 | 85 | 78 | 325
Age, Continuous [Mean (Full Range); unit: years] | 42.1 [24 to 55] | 40.8 [23 to 55] | 42.7 [21 to 55] | 40.9 [19 to 55] | 41.6 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 25 | 23 | 94
  Male | 60 | 56 | 60 | 55 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 9 | 15 | 41
  Not Hispanic or Latino | 72 | 72 | 76 | 63 | 283
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 1 | 1 | 0 | 4
  Race: Asian | 2 | 4 | 1 | 2 | 9
  Race: Black or African American | 49 | 57 | 57 | 47 | 210
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
  Race: White | 23 | 18 | 23 | 26 | 90
  Race: Other | 4 | 1 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 12
Description: PANSS measures symptom severity in participants with schizophrenia. PANSS includes 30 items (7 items for positive symptoms, 7 items for negative symptoms, and 16 items for general psychopathology symptoms), and each item is rated with 1 to 7 points. The PANSS is scored by summation of ratings across items such that the score ranges are 7 to 49 for each of the Positive and Negative Scales and 16 to 112 for the General Psychopathology Scale. The PANSS total score is a sum of scores from all the 30 items and the scores range from 30 to 210, where a higher score represents more severe symptoms, and lower scores represent a better quality of life in participants with schizophrenia. A negative change from baseline indicates low severity of symptoms.
Time Frame: Baseline, Week 12
Population: Efficacy population included all participants who received the study medication and had at least one available post-baseline PANSS assessment. 'Number of participants analyzed' indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-692 1 Gram QD | CTP-692 2 Grams QD | CTP-692 4 Grams QD
Number analyzed (Participants) | 80 | 81 | 83 | 77
score on a scale
  Baseline | 82.1 (8.2) | 81.2 (8.0) | 81.6 (7.8) | 82.9 (8.6)
  Change From Baseline at Week 12: number analyzed (Participants) | 63 | 54 | 63 | 65
  Change From Baseline at Week 12 | -14.1 (10.4) | -15.9 (10.3) | -12.2 (10.3) | -11.0 (10.6)
Statistical Analysis 1: Comparison: Placebo vs CTP-692 1 Gram QD; Test type: Superiority; p = 0.6003, Mixed model repeated measures (MMRM); MMRM included fixed effects of treatment group, analysis visit, treatment-by-visit interaction, and a baseline-by-visit interaction; Least Square (LS) Mean Difference = -0.9, 95% CI 2-sided [-4.5 to 2.6], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: Placebo vs CTP-692 2 Grams QD; Test type: Superiority; p = 0.3920, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.5, 95% CI 2-sided [-2.0 to 5.0], Standard Error of Mean 1.8
Statistical Analysis 3: Comparison: Placebo vs CTP-692 4 Grams QD; Test type: Superiority; p = 0.1444, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.6, 95% CI 2-sided [-0.9 to 6.0], Standard Error of Mean 1.8

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 12
Description: The CGI-S rating scale is a commonly used measure of symptom severity and treatment response. CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment and the score ranges from 1 to 7: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. A higher score represents more severe symptoms. A negative change from baseline indicates low severity of symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-692 1 Gram QD | CTP-692 2 Grams QD | CTP-692 4 Grams QD
Number analyzed (Participants) | 80 | 81 | 83 | 77
score on a scale
  Baseline | 4.2 (0.5) | 4.1 (0.5) | 4.1 (0.5) | 4.2 (0.6)
  Change From Baseline at Week 12: number analyzed (Participants) | 63 | 54 | 63 | 65
  Change From Baseline at Week 12 | -0.8 (0.8) | -0.8 (0.9) | -0.5 (0.7) | -0.5 (0.7)
Statistical Analysis 1: Comparison: Placebo vs CTP-692 1 Gram QD; Test type: Superiority; p = 0.8065, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs CTP-692 2 Grams QD; Test type: Superiority; p = 0.2121, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.4], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Placebo vs CTP-692 4 Grams QD; Test type: Superiority; p = 0.0264, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [0.0 to 0.5], Standard Error of Mean 0.1

3. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Scale at Week 12
Description: PSP scale is a measure of the personal and social functioning of participants with psychiatric disorders within four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. Each domain was assessed on a 6-point scale: 1 = absent, 2 = mild, 3 = manifest, 4 = marked, 5 = severe, and 6 = very severe. The final global score is defined according to a summary instruction table converting four domain scores into a single, overall rating from 1 to 100: 71 to 100 represent mild degree of difficulty; 31 to 70 represent varying degrees of disability, and 1 to 30 represent functioning so poorly as to require intensive supervision. Higher scores represent better personal and social function. A positive change from baseline indicates better personal and social function.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CTP-692 1 Gram QD | CTP-692 2 Grams QD | CTP-692 4 Grams QD
Number analyzed (Participants) | 80 | 81 | 83 | 77
score on a scale
  Baseline | 57.5 (10.0) | 58.7 (8.9) | 58.4 (9.8) | 58.0 (9.2)
  Change From Baseline at Week 12: number analyzed (Participants) | 63 | 54 | 63 | 65
  Change From Baseline at Week 12 | 4.3 (8.6) | 4.6 (9.1) | 3.7 (7.4) | 2.3 (8.3)
Statistical Analysis 1: Comparison: Placebo vs CTP-692 1 Gram QD; Test type: Superiority; p = 0.6101, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [-2.1 to 3.5], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: Placebo vs CTP-692 2 Grams QD; Test type: Superiority; p = 0.6237, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-3.4 to 2.1], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: Placebo vs CTP-692 4 Grams QD; Test type: Superiority; p = 0.1764, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-4.6 to 0.8], Standard Error of Mean 1.4

ADVERSE EVENTS:
Time Frame: All-cause mortality: Screening up to the last follow-up visit (approximately 18 weeks); Adverse events: From the first dose of study medication up to the last follow-up visit (approximately 13 weeks)
Description: All-cause mortality: All randomized participants included all participants who were randomized in the study.
  Adverse events: Safety population included all participants who received at least one dose of study medication.
Arm/Group | Placebo | CTP-692 1 Gram QD | CTP-692 2 Grams QD | CTP-692 4 Grams QD
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81 | 0/85 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/81 | 1/81 | 0/85 | 1/78
Other Adverse Events (participants affected / at risk) | 3/81 | 5/81 | 6/85 | 7/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | CTP-692 1 Gram QD (N=81) | CTP-692 2 Grams QD (N=85) | CTP-692 4 Grams QD (N=78)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | CTP-692 1 Gram QD (N=81) | CTP-692 2 Grams QD (N=85) | CTP-692 4 Grams QD (N=78)
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 4
Headache (Nervous system disorders) | 2 | 4 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wants to publish study data or results, the publication or presentation must be provided to Concert for review at least 60 days in advance. If Concert needs to file a patent application prior to publication, the publication can be delayed up to 90 days from Sponsor providing notice to the investigator of such need.

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT04158687/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT04158687/SAP_001.pdf